CLINICAL TRIAL: NCT06074003
Title: Does Biological Sex Influence Insulin Sensitivity and Muscle Metabolism Following High-intensity Interval Exercise?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Jenna Gillen, Assistant Professor, University of Toronto
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 44435
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2024-12

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Females (Experimental): Female participant group
  Interventions: Other: Seated Rest (Non-exercise control); Other: High-intensity interval exercise
- Males (Experimental): Male participant group
  Interventions: Other: Seated Rest (Non-exercise control); Other: High-intensity interval exercise

INTERVENTIONS:
Other: Seated Rest (Non-exercise control) — Sitting for 30 minutes
Other: High-intensity interval exercise — Performing a single session of high-intensity interval exercise on a cycle ergometer

SUMMARY:
High-intensity interval exercise (HIIE) is a type of exercise that involves alternating periods of intense exercise with periods of rest. HIIE has been shown to improve many aspects of cardiovascular and metabolic health in a time-efficient manner (e.g., only 20 minutes per exercise session). An important health benefit of exercise is improved blood sugar control, which can help reduce the risk of metabolic diseases like type 2 diabetes. A single session of HIIE has been shown to improve blood sugar in males, but it is unknown if females achieve the same health benefit. It is also not fully understood how exercise improves blood sugar in males and females. Therefore, the purpose of this project is 1) to determine if a single session of HIIE improves blood sugar control in males and females, and 2) to evaluate if changes in skeletal muscle can explain the beneficial effects of HIIE on blood sugar.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine if biological sex influences the effects of high-intensity interval exercise (HIIE) on insulin sensitivity and muscle mechanisms. The investigators will measure insulin sensitivity and muscle outcomes of participants on two separate occasions: 1) Following 30 minutes of sitting in the lab; and 2) Following a single session of HIIE on a stationary bike. Insulin sensitivity will be measured by taking blood samples after participants consume a sugary drink. Muscle outcomes will be measured by taking a small amount of muscle from the vastus lateralis (thigh) muscle. Groups of male and female participants will be recruited and tested using best practice guidelines for sex-based comparisons of exercise responses.

The study will advance knowledge regarding the potential for biological sex to influence the metabolic responses high-intensity exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 yrs
* VO2peak considered recreationally active as defined as 'fair' or 'good' (males: 41.6- 50.5ml/kg/min; females: 35-41.9 ml/kg/min) based on Canadian Society for Exercise Physiology (CSEP) normative fitness values.
* BMI between 18-27 kg/m2
* 1-3 structured exercise sessions/week, and not training for any specific sport
* Weight stable (within ± 2kg for at least 6 months)
* Eumenorrheic (female only), defined as menstrual cycle lengths ≥ 21 days and ≤ 35 days resulting in 9 or more consecutive periods per year)
* Non-smoker

Exclusion Criteria:

* Diagnosed with cardiovascular or metabolic disease, hyper- or hypogonadism, and/or polycystic ovarian syndrome (PCOS)
* The use of medication for managing blood glucose or lipid metabolism
* Current use of oral contraceptives or use within the last 3 months
* Irregular menstrual cycles (<21 days or >35 days)
* Pregnant, lactating, or menopausal
* Recreational smoking of any kind
* Inability to perform the study exercise protocols or follow the pre-trial dietary or physical activity controls
* Taking medications affecting substrate metabolism (corticosteroids or nSAIDs)
* Actively engaging in a low-carbohydrate diet (e.g., ketogenic, Atkins)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-06-26 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Insulin area under the curve | 3 hours
  Insulin area under the curve measured during glucose tolerance test

SECONDARY OUTCOMES:
Glucose area under the curve | 3 hours
  Glucose area under the curve measured during glucose tolerance test
Mean insulin concentration | 3 hours
  Mean insulin concentration measured during glucose tolerance test
Mean glucose concentration | 3 hours
  Mean glucose concentration measured during glucose tolerance test
Peak insulin concentration | 3 hours
  Peak insulin concentration measured during the glucose tolerance test
Peak glucose concentration | 3 hours
  Peak insulin concentration measured during the glucose tolerance test
Insulin:glucose ratio | 3 hours
  Insulin to glucose ration measured during the glucose tolerance test
Postprandial glucose oxidation | 3 hours
  Postprandial glucose oxidation measured with a metabolic tracer
Skeletal muscle glycogen content | immediately before and after exercise
  Muscle glycogen use during exercise
Skeletal muscle contractile signaling protein content | immediately before and after exercise
  Measured via western blotting
Skeletal muscle insulin signaling | 1hr into glucose tolerance test
  Measured via western blotting
Mitochondrial gene expression | Change from pre-exercise to 3hr post-exercise
  Measured via Reverse transcription polymerase chain reaction
Muscle protein synthesis rates | 3hr post-exercise
  Muscle protein synthesis rates assessed by incorporation of oral stable isotope tracer following exercise
Local muscle oxygenation | During exercise
  Muscle oxygenation (vastus lateralis) assessed with near-infrared spectroscopy (NIRS)
Local muscle oxygenation | Pre-exercise, immediately post-exercise and 2 hrs post-exercise
  Muscle oxygenation (vastus lateralis) assessed with NIRS during and following thigh cuff inflation

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Estafanos, MSc, Study Director — University of Toronto
Locations (1):
- Goldring Centre for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No